CLINICAL TRIAL: NCT00900991
Title: Safety and Immunogenicity of a Split-Virion Pandemic Influenza A (H5N1) Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-sPanFlu-2002
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Influenza
Keywords: Pandemic Influenza A Vaccine; Immunogenictiy; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 ug (Experimental): 10 microgram per dose
  Interventions: Biological: split-virion pandemic influenza vaccine (H5N1 strain NIBRG-14)
- 15 ug (Experimental): 15 microgram per dose
  Interventions: Biological: split-virion pandemic influenza vaccine (H5N1 strain NIBRG-14)

INTERVENTIONS:
Biological: split-virion pandemic influenza vaccine (H5N1 strain NIBRG-14)

SUMMARY:
A single center, stratified, randomized and double-blind phase II clinical trial was conducted in children to evaluate the safety and immunogenicity of an split-virion pandemic influenza A vaccine (H5N1).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 3-11 years old
* Be able to show legal identity card for the sake of recruitment
* Volunteers or their parents are able to understand and sign the informed consent
* Do not participate in other clinical trial

Exclusion Criteria:

* Any history of allergic reactions
* Autoimmune disease or immunodeficiency
* Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
* Diabetes mellitus (type I or II), with the exception of gestational diabetes
* History of thyroidectomy or thyroid disease that required medication within the past 12 months
* Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
* Hypertension that was not well controlled by medication or the blood pressure is more than 145/95 mmHg at enrollment
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
* Seizure disorder other than:

  1. Febrile seizures under the age of two years old
  2. Seizures secondary to alcohol withdrawal more than 3 years ago, or
  3. A singular seizure not requiring treatment within the last 3 years
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* Guillain-Barre Syndrome
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
* History of any blood products administration within 3 months before the dosing
* Administration of any other investigational research agents within 30 days before the dosing
* Administration of any live attenuated vaccine within 30 days before the dosing
* Administration of subunit or inactivated vaccines, e.g. pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
* Be receiving anti-TB prophylaxis or therapy currently
* Axillary temperature > 37.0 centigrade at the time of dosing
* Psychiatric condition that precludes compliance with the protocol:

  1. Past or present psychoses
  2. Past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years
  3. Disorder requiring lithium
  4. Suicidal ideation occurring within five years prior to enrollment
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

PRIMARY OUTCOMES:
HI antibody and Neutralization antibody

SECONDARY OUTCOMES:
Adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Centers for Diseases Control and Prevention, Beijing, China